CLINICAL TRIAL: NCT00543465
Title: 12-Week No-Rofecoxib Plus Aspirin Endoscopy Study (0782-003)
Status: Terminated | Phase: Phase 2 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 0782-003; 2007_636
Record Dates: First submitted 2007-10-05; First posted 2007-10-15 (Estimated); Last update posted 2015-06-02 (Estimated); Status verified 2015-06

CONDITIONS: Arthritis, Rheumatoid; Osteoarthritis
MeSH Terms: conditions — Arthritis, Rheumatoid; Osteoarthritis

STUDY DESIGN:
Who Masked: Participant, Investigator

INTERVENTIONS:
Drug: MK0782

SUMMARY:
This study will look at the incidence of gastric and/or duodenal ulcers in patients with osteoarthritis or rheumatoid arthritis in four different treatment groups (a) MK0782 21 mg plus enteric-coated aspirin, (b) MK0782 42 mg plus enteric-coated aspirin, (c) celecoxib 200 mg plus enteric-coated aspirin, and enteric-coated aspiring alone.

This is an early phase trial and some specific protocol information is in progress and not publicly available at this time. (Full information is available to trial participants).

ELIGIBILITY:
Inclusion Criteria:

* Has osteoarthritis or rheumatoid arthritis for at least 6 months prior to start of study
* Osteoarthritis (OA): must have diagnosis of OA in knee, hip, hand or spine

Patient is not on chronic aspirin therapy (taking aspirin at any dose, on a daily basis, for a minimum of 4 weeks prior to Visit 2 for any medical condition

* Must be willing to limit alcohol use to no more than 2 drinks per day
* Avoid strenuous physical activity

Exclusion Criteria:

* Mentally or legally incapacitated
* Has systemic lupus erythematosus, Paget's disease
* Has a history of esophageal, gastric biliary, or small intestine surgery (hiatal surgeries and any GI surgery that causes clinical malabsorption or delayed gastric emptying
* Has uncontrolled hypertension
* Has uncontrolled diabetes
* Has had heart attack, unstable angina, coronary angioplasty, stent placement, coronary artery bypass grafting in the last 6 months
* Has congestive heart failure
* Has had active liver disease within the last 2 years

Min Age: 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 49 (Actual)
Dates: Start 2004-08; Primary Completion 2004-11 (Actual); Study Completion 2004-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Merck Sharp & Dohme LLC